CLINICAL TRIAL: NCT03840031
Title: SASHA-II Iron Bioavailability From Iron-biofortified Orange Fleshed Sweet Potato in Malawian Women Between 18-35 Years
Brief Title: Iron Bioavailability From Biofortified Orange-fleshed Sweet Potato
Acronym: SASHA-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Malawi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: SASHA-II
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia
Keywords: Biofortification; Orange fleshed sweet potato; Stable isotope studies
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: Each woman consumes both Orange Fleshed Sweet Potato varieties
Who Masked: Participant
Masking Description: Participant is blinded, meal option A --> B or B --> A based on investigator randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orange Fleshed Sweet Potato High Iron (Experimental): Meal sequence B, OFSP High Fe
  Interventions: Other: High Fe OFSP meal labelled with Fe-58
- Orange Fleshed Sweet Potato Control (Active Comparator): Meal sequence A, OFSP control
  Interventions: Other: Control OFSP meal labelled with Fe-57

INTERVENTIONS:
Other: High Fe OFSP meal labelled with Fe-58 — 400 gram steamed, mashed OFSP high Fe with 0.33 mg FeSO4-58 daily for 10 days
  Arms: Orange Fleshed Sweet Potato High Iron
Other: Control OFSP meal labelled with Fe-57 — 400 gram steamed, mashed OFSP control with 0.33 mg FeSO5-57 daily for 10 days
  Arms: Orange Fleshed Sweet Potato Control

SUMMARY:
To combat iron deficiency in Low and Middle-Income Countries, sustainable food-based solutions have to be implemented to serve populations, not only individuals. One solution is the introduction of iron biofortified staple crops on market level. Before market level introduction, the bioavailability of iron in the new biofortified Orange Fleshed Sweet Potato (OFSP) breed needs to be assessed. In this study the investigator compares the fractional and total iron absorption after extrinsic stable isotope labelling of the new biofortified high iron OFSP variety and a normal market level OFSP variety. The study is conducted in Malawian women of reproductive age with marginal iron status.

DETAILED DESCRIPTION:
The 25 women enrolled will consume test meals consisting of 400g steamed and mashed high iron sweet potatoes labelled with Fe-58 daily for a period of 10 days and will then switch to the test meals consisting of 400g steamed and mashed control sweet potatoes labelled with Fe-57 for a period of 10 days. The order of test meal type is random. A baseline blood sample will be taken on the first meal feeding day prior to consumption of any test meals, on study day 26 (14 days after completion of the first test meal period) and on Day 40 (14 days after completion of the second test meal period). Erythrocyte incorporation of the stable isotope labels will be measured in these blood samples using an ICPMS and will be used to calculate fractional and total iron absorption from the two different type of test meals.

ELIGIBILITY:
Inclusion Criteria:

1. Woman aged 18-35 years old
2. low/marginal iron status respectively evidenced by one of the following criteria: PF ≤ 25 µg/L
3. Normal BMI for age (18.5-25.0 kg/m2)
4. Weight less than 65 kg. A maximum weight limitation is needed since the stable isotope portions are based on body weight. We want to give equal amounts of stable isotopes to each study participant and therefore need to standardize body weight.
5. Living in a study radius of 30 km from the meal distribution/ health centre side
6. Willing and able to commute to the set meal distribution/ health centre side
7. Able to understand and to sign* written concept prior to trial entry
8. Informed consent signed * Signing of informed consent by either autograph or finger print.

Exclusion Criteria:

1. Severe anaemia Hb <80 g/l
2. High infection rate based on CRP > 5 mg/L
3. Any known chronic diseases
4. Relevant digestive (intestinal, gastric, hepatic or pancreatic), renal, metabolic disease, as determined by the screening visit and by self-report from the subjects.
5. Diagnosed food allergy.
6. Pregnancy (urine test during screening
7. Lactation.
8. History of cancer within the past year, from self-report by the woman or as obtained from her health passport
9. Any medication or supplement which may impact erythrocytes, Hb or haematocrit (to the opinion of the investigator).
10. Iron supplementation therapy or perfusion in the last three months
11. Significant blood losses over the past 6 months (i.e. trauma, major surgery, blood donation or other cause influencing blood volume to be investigated by the PI)
12. Have a high alcohol consumption (more than 2 drinks/day).
13. Consumption of illicit drugs based on reported use (based on anamnesis only).
14. Subject having a hierarchical link with the investigator or co-investigators.
15. Fever (body temperature >37.5 °C), on day 1 of the feeding scheme
16. Subject who cannot be expected to comply with treatment (malaria or helminths) or study procedure.
17. Currently participating or having participated in another clinical trial during the past month prior to the beginning of this study.
18. Enrolment in any (micronutrient) food program
19. Subjects not willing and/or not able to comply with scheduled visits and the requirements of the study protocol.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Based on health passport or birth certificate.
Enrollment: 25 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption from both Orange Fleshed Sweet Potato varieties | Measured 2 weeks after completion of feeding day sequence. Sequence consist of 2 times 10 feeding days.
  Proportion of stable isotope administered with test meals that has been incorporate into erythrocytes 14 days after completion of specific test meal feeding period
Total iron absorption from both Orange Fleshed Sweet Potato varieties | Measured 2 weeks after completion of feeding day sequence. Sequence consist of 2 times 10 feeding days.
  Amount of iron absorbed (mg) from the labelled test meals

SECONDARY OUTCOMES:
Concentration of plasma ferritin level | screening (-1), baseline (day 1), last test meal consumption (day 26) and 14 days after last test meal consumption (day 40)
  Iron status marker
Concentration of plasma CRP level | screening (-1), baseline (day 1), last test meal consumption (day 26) and 14 days after last test meal consumption (day 40)
  Inflammation status marker

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, Prof., Principal Investigator — Swiss Federal Institute of Technology
Locations (2):
- Training and Research Unit of Excellence, University of Malawi, Zomba, Malawi
- Swiss Federal Institute of Technology, Laboratory of Human Nutrition, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jongstra R, Mwangi MN, Burgos G, Zeder C, Low JW, Mzembe G, Liria R, Penny M, Andrade MI, Fairweather-Tait S, Zum Felde T, Campos H, Phiri KS, Zimmermann MB, Wegmuller R. Iron Absorption from Iron-Biofortified Sweetpotato Is Higher Than Regular Sweetpotato in Malawian Women while Iron Absorption from Regular and Iron-Biofortified Potatoes Is High in Peruvian Women. J Nutr. 2020 Dec 10;150(12):3094-3102. doi: 10.1093/jn/nxaa267. PMID 33188398